CLINICAL TRIAL: NCT04537897
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of BI 474121 in Young and Elderly Healthy Male and Female Subjects (Double-blind, Randomised, Placebo-controlled, Parallel Group Design) and Evaluation of Midazolam Interaction in Young Healthy Male and Female Subjects (Nested, Open, Fixed-sequence, Intra-individual Comparison)
Brief Title: A Study in Healthy Men and Women Who Are Either Between 18 - 45 Years or Between 65 - 80 Years to Test How Different Doses of BI 474121 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1411-0002; 2020-001003-17 (EudraCT Number)
Record Dates: First submitted 2020-08-31; First posted 2020-09-03 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- BI 474121 2.5mg (Part A) (Experimental): Young participants administered 1 tablet of 2.5 milligrams (mg) BI 474121 orally once daily over a treatment period of 14 days.
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily.
  Interventions: Drug: BI 474121; Drug: Midazolam
- BI 474121 5mg (Part A) (Experimental): Young participants administered 2 tablets of 2.5 mg BI 474121 orally once daily (daily dose: 5 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days.
  Interventions: Drug: BI 474121
- BI 474121 10mg (Part A) (Experimental): Young participants administered 1 tablet of 10 milligrams (mg) BI 474121 orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days.
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: BI 474121; Drug: Midazolam
- BI 474121 20mg (Part A) (Experimental): Young participants administered 2 tablets of 10 milligrams (mg) BI 474121 orally once daily (daily dose: 20 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days.
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: BI 474121; Drug: Midazolam
- BI 474121 30mg (Part A) (Experimental): Young participants administered 3 tablets of 10 milligrams (mg) BI 474121 orally once daily (daily dose: 30 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days.
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: BI 474121; Drug: Midazolam
- Placebo (Part A) (Placebo Comparator): Young participants administered matching placebo to part A once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days.
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) for placebo participants matched to 2.5mg BI, 10mg BI, 20mg BI, and 30mg BI groups.
  Interventions: Drug: BI 474121; Drug: Midazolam; Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Elderly participants administered matching placebo to part B once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days
  Interventions: Drug: Placebo
- BI 474121 5mg (Part B) (Experimental): Elderly participants administered 2 tablets of 2.5 mg BI 474121 orally once daily (daily dose: 5 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days.
  Interventions: Drug: BI 474121
- BI 474121 10mg (Part B) (Experimental): Elderly participants administered 1 tablet of 10 milligrams (mg) BI 474121 orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days.
  Interventions: Drug: BI 474121

INTERVENTIONS:
Drug: BI 474121 — BI474121
  Arms: BI 474121 10mg (Part A); BI 474121 10mg (Part B); BI 474121 2.5mg (Part A); BI 474121 20mg (Part A); BI 474121 30mg (Part A); BI 474121 5mg (Part A); BI 474121 5mg (Part B); Placebo (Part A)
Drug: Midazolam — Midazolam
  Arms: BI 474121 10mg (Part A); BI 474121 2.5mg (Part A); BI 474121 20mg (Part A); BI 474121 30mg (Part A); Placebo (Part A)
Drug: Placebo — Placebo
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main objectives of this trial are to investigate safety and tolerability of BI 474121 in healthy male and female young and elderly subjects following oral administration of multiple rising doses per day over 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 45 years (inclusive) for young or 65 to 80 years (inclusive) for elderly healthy volunteers
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mm Hg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* A positive Poly-chain reaction (PCR) test for SARS-CoV-2 and clinical symptoms suggestive for this disease at screening or on Day -3
* Further exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial investigated the safety, tolerability, and pharmacokinetics (PK) of BI 474121 in healthy male and female young and elderly subjects following oral administration of multiple rising doses per day over 14 days and to investigate the effect of BI 474121 on the PK of midazolam, given as an oral microdose.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all patients as required.
Groups:
- Placebo (Part A): Young participants administered matching placebo to 2.5 milligram (mg) and 10 mg tablets once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days (Day 1 - Day 14).
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) for placebo participants matched to 2.5mg BI, 10mg BI, 20mg BI, and 30mg BI groups.
- BI 474121 2.5mg (Part A): Young participants administered 1 tablet of 2.5 milligrams (mg) BI 474121 orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days (Day 1 - Day 14).
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
- BI 474121 5mg (Part A): Young participants administered 2 tablets of 2.5 mg BI 474121 orally once daily (daily dose: 5 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days (Day 1 - Day 14).
- BI 474121 10mg (Part A): Young participants administered 1 tablet of 10 milligrams (mg) BI 474121 orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days (Day 1 - Day 14).
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
- BI 474121 20mg (Part A): Young participants administered 2 tablets of 10 milligrams (mg) BI 474121 orally once daily (daily dose: 20 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days (Day 1 - Day 14).
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
- BI 474121 30mg (Part A): Young participants administered 3 tablets of 10 milligrams (mg) BI 474121 orally once daily (daily dose: 30 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days (Day 1 - Day 14).
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h).
- Placebo (Part B): Elderly participants administered matching placebo to 2.5 mg and 10 mg tablets once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days (Day 1 - Day 14).
- BI 474121 5mg (Part B): Elderly participants administered 2 tablets of 2.5 mg BI 474121 orally once daily (daily dose: 5 mg) with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days (Day 1 - Day 14).
- BI 474121 10mg (Part B): Elderly participants administered 1 tablet of 10 milligrams (mg) BI 474121 orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days (Day 1 - Day 14).
Period: Overall Study
Arm/Group | Placebo (Part A) | BI 474121 2.5mg (Part A) | BI 474121 5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part B) | BI 474121 5mg (Part B) | BI 474121 10mg (Part B)
Started | 10 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8
Completed ("Completed" = not prematurely discontinued from trial medication.) | 10 | 7 | 8 | 7 | 8 | 8 | 3 | 8 | 8
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Other than listed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | BI 474121 2.5mg (Part A) | BI 474121 5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part B) | BI 474121 5mg (Part B) | BI 474121 10mg (Part B) | Total
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (5.3) | 35.4 (8.9) | 31.4 (9.5) | 31.3 (7.1) | 32.4 (7.7) | 29.3 (5.7) | 66.5 (2.4) | 70.8 (4.7) | 72.3 (5.3) | 42.4 (19.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 3 | 5 | 5 | 2 | 1 | 4 | 29
  Male | 8 | 5 | 4 | 5 | 3 | 3 | 2 | 7 | 4 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 10 | 7 | 8 | 8 | 8 | 7 | 4 | 7 | 8 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  White | 8 | 8 | 7 | 7 | 8 | 8 | 4 | 8 | 8 | 66
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events
Description: Percentage of participants with drug-related adverse events is reported. Medical judgment were used to determine the relationship between study medication and the adverse events, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.
Time Frame: For Midazolam: From first dose of midazolam (on Day -1) until first dose of BI 474121/Placebo, up to 1 day. Other groups: From first dose of BI 474121/Placebo until last dose+7 days of residual effect period, up to 21 days.
Population: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug.
Measure: Number; unit: Percentage of participants
Groups:
- Midazolam: 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) on Day -1 for young participants assigned to 2.5mg, 10,mg, 20mg, and 30mg BI/Placebo groups.
Arm/Group | Placebo (Part A) | BI 474121 2.5mg (Part A) | BI 474121 5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part B) | BI 474121 5mg (Part B) | BI 474121 10mg (Part B) | Midazolam
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8 | 40
Percentage of participants | 40.0 | 75.0 | 50.0 | 75.0 | 87.5 | 100.0 | 25.0 | 25.0 | 50.0 | 12.5

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 474121 in Plasma From 0 to 24h (AUC0-24) After First Dose
Description: The area under the concentration-time curve of BI 474121 in plasma from 0 to 24h (AUC0-24) after first dose is reported.
Time Frame: Within 1 hour (h) before and at 15 minutes (min), 30min, 1h, 1h30min, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 23h45min after first dose of BI 474121.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the treated set who provided at least 1 PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Only participants with non-missing results were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomole / Liter (h*nmol/L)
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | BI 474121 5mg (Part B) | BI 474121 10mg (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8 | 8
hour * nanomole / Liter (h*nmol/L) | 230 (20.9) | 486 (23.1) | 862 (19.1) | 1650 (23.4) | 2430 (20.0) | 410 (34.2) | 891 (13.7)

3. Secondary Outcome: Maximum Measured Concentration of BI 474121 in Plasma (Cmax) After First Dose
Description: The maximum measured concentration of BI 474121 in plasma (Cmax) after first dose is reported.
Time Frame: as for outcome 2
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the treated set who provided at least 1 PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole / Liter (nmol/L)
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | BI 474121 5mg (Part B) | BI 474121 10mg (Part B)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
nanomole / Liter (nmol/L) | 22.6 (29.7) | 43.9 (19.8) | 82.4 (25.9) | 167 (33.2) | 229 (20.2) | 44.3 (37.7) | 89.4 (15.0)

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 474121 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss)
Description: The area under the concentration-time curve of BI 474121 in plasma at steady state over a uniform dosing interval τ (dosing interval = 24 hours) (AUCτ,ss) is reported.
Time Frame: Within 15 minutes (min) before and at 15 min, 30min, 1hour (h), 1h30min, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h after administration of BI 474121 on Day 14.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomole / Liter (h*nmol/L)
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | BI 474121 5mg (Part B) | BI 474121 10mg (Part B)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 8 | 8 | 8
hour * nanomole / Liter (h*nmol/L) | 471 (28.3) | 797 (31.6) | 1280 (25.1) | 2870 (26.4) | 4350 (27.4) | 764 (39.4) | 1640 (19.7)

5. Secondary Outcome: Maximum Measured Concentration of BI 474121 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss)
Description: The maximum measured concentration of BI 474121 in plasma at steady state over a uniform dosing interval τ (dosing interval = 24 hours) (Cmax,ss) is reported.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole / Liter (nmol/L)
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | BI 474121 5mg (Part B) | BI 474121 10mg (Part B)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 8 | 8 | 8
nanomole / Liter (nmol/L) | 40.1 (26.3) | 67.8 (22.2) | 113 (19.6) | 249 (23.9) | 385 (26.8) | 60.6 (40.0) | 142 (12.2)

6. Secondary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Cmax) - Day -1
Description: The maximum measured concentration of Midazolam in plasma (Cmax) on Day -1 is reported.
Time Frame: Within 1 hour (h) 30 minutes (min) before and at 15min, 30min, 1h, 1h30min, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 23h after the administration of Midazolam on Day -1.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole / Liter (pmol/L)
Groups:
- Placebo (Part A) (Midazolam): Young participants administered matching placebo to part A (matching to 2.5mg, 10mg, 20mg, and 30mg BI groups) once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) over a treatment period of 14 days.
  On Day -1, 1, and 14, 75 micrograms (μg) of midazolam for injection used as oral solution were administered orally once daily with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h) for placebo participants matched to 2.5mg BI, 10mg BI, 20mg BI, and 30mg BI groups.
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part A) (Midazolam)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
picomole / Liter (pmol/L) | 980 (34.8) | 747 (20.2) | 1460 (37.4) | 981 (32.7) | 901 (28.8)

7. Secondary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Cmax) - Day 1
Description: The Maximum measured concentration of Midazolam in plasma (Cmax) on Day 1 is reported.
Time Frame: Within 1 hour (h) before and at 15 minutes (min), 30min, 1h, 1h30min, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 23h45min after administration of Midazolam on Day 1.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole / Liter (pmol/L)
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part A) (Midazolam)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
picomole / Liter (pmol/L) | 1090 (44.7) | 913 (35.2) | 1210 (36.3) | 934 (44.8) | 987 (31.3)

8. Secondary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Cmax) - Day 14
Description: The Maximum measured concentration of Midazolam in plasma (Cmax) on Day 14 is reported.
Time Frame: Within 15 minutes (min) before and at 15min, 30min, 1hour (h), 1h30min, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h after administration of Midazolam on Day 14.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole / Liter (pmol/L)
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part A) (Midazolam)
Number analyzed (Participants) | 7 | 7 | 8 | 8 | 8
picomole / Liter (pmol/L) | 1250 (42.0) | 1010 (28.2) | 1160 (45.4) | 1090 (51.9) | 931 (31.3)

9. Secondary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) - Day -1
Description: The area under the concentration-time curve of Midazolam in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) on Day -1 is reported.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * picomole / Liter (h * pmol/L)
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part A) (Midazolam)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
hour * picomole / Liter (h * pmol/L) | 2830 (59.8) | 1920 (27.2) | 3080 (30.8) | 2610 (56.9) | 2350 (38.5)

10. Secondary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) - Day 1
Description: The Area under the concentration-time curve of Midazolam in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) on Day 1 is reported.
Time Frame: as for outcome 7
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * picomole / Liter (h * pmol/L)
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part A) (Midazolam)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
hour * picomole / Liter (h * pmol/L) | 2760 (58.3) | 2020 (25.8) | 2720 (31.4) | 2290 (85.8) | 2360 (40.7)

11. Secondary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) - Day 14
Description: The Area under the concentration-time curve of Midazolam in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) on Day 14 is reported.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * picomole / Liter (h * pmol/L)
Arm/Group | BI 474121 2.5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part A) (Midazolam)
Number analyzed (Participants) | 7 | 7 | 8 | 8 | 8
hour * picomole / Liter (h * pmol/L) | 3570 (44.7) | 2130 (30.6) | 2710 (38.0) | 2390 (74.2) | 2570 (37.6)

ADVERSE EVENTS:
Time Frame: For Midazolam: From first dose of midazolam (on Day -1) until first dose of BI 474121/Placebo, up to 1 day. Other groups: From first dose of BI 474121/Placebo until last dose+7 days of residual effect period, up to 21 days.
Description: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug.
Arm/Group | Placebo (Part A) | BI 474121 2.5mg (Part A) | BI 474121 5mg (Part A) | BI 474121 10mg (Part A) | BI 474121 20mg (Part A) | BI 474121 30mg (Part A) | Placebo (Part B) | BI 474121 5mg (Part B) | BI 474121 10mg (Part B) | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/4 | 0/8 | 0/8 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/4 | 0/8 | 0/8 | 0/40
Other Adverse Events (participants affected / at risk) | 5/10 | 7/8 | 4/8 | 6/8 | 7/8 | 8/8 | 1/4 | 4/8 | 5/8 | 6/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A) (N=10) | BI 474121 2.5mg (Part A) (N=8) | BI 474121 5mg (Part A) (N=8) | BI 474121 10mg (Part A) (N=8) | BI 474121 20mg (Part A) (N=8) | BI 474121 30mg (Part A) (N=8) | Placebo (Part B) (N=4) | BI 474121 5mg (Part B) (N=8) | BI 474121 10mg (Part B) (N=8) | Midazolam (N=40)
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 4
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site thrombosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure orthostatic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glutamate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myoglobin blood increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic heart rate response increased (Investigations) | 2 | 4 | 3 | 4 | 6 | 4 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 0
Dizziness exertional (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug withdrawal headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 1 | 5 | 2 | 1 | 1 | 1 | 2
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Impulsive behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT04537897/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT04537897/SAP_001.pdf